CLINICAL TRIAL: NCT01713855
Title: Vaccine Response After Rituximab for Chronic, Severe Idiopathic Thrombocytopenic Purpura (ITP)
Brief Title: Vaccine Response After Rituximab for Chronic, Severe Idiopathic Thrombocytopenic Purpura
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neufeld, Ellis J, MD, PhD (Individual)
Collaborators: Terrana ITP Research Fund (Other)
Responsible Party: Ellis J. Neufeld, MD, PhD, Children's Hospital Boston
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: CHB 04-10-143
Record Dates: First submitted 2012-10-18; First posted 2012-10-25 (Estimated); Last update posted 2012-10-25 (Estimated); Status verified 2012-10

CONDITIONS: Idiopathic Thrombocytopenic Purpura; Immune Thrombocytopenic Purpura
Keywords: ITP; Rituximab; Vaccine; Immune Reconstitution
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Inactivated Trivalent Influenza vaccine

SUMMARY:
The purpose of this study is to determine how children with a history of severe, chronic Idiopathic Thrombocytopenic Purpura (ITP) who were treated with rituximab might respond to vaccines. Eligible patients are previously or currently enrolled in a study entitled "Open Label, Phase I/II Trial of Rituximab for Chronic, Severe Idiopathic Thrombocytopenic Purpura in Children and Adolescents" and have decided to obtain an inactivated influenza vaccination. These patients will be invited to provide one blood sample prior to vaccination and a second sample following vaccination to quantify immune response to vaccination.

DETAILED DESCRIPTION:
The purpose of this ancillary, pilot-phase study is to determine how children with a history of severe, chronic ITP who were treated with rituximab might respond to vaccines. Eligible patients are previously or currently enrolled in a study entitled "Open Label, Phase I/II Trial of Rituximab for Chronic, Severe Idiopathic Thrombocytopenic Purpura in Children and Adolescents" (CHB 02-12-160) and have decided to obtain the trivalent, inactivated influenza vaccination. These patients will be invited to provide one blood sample prior to vaccination and a second sample 4-8 weeks after vaccination to quantify immune response to vaccination. Additionally, if patients are scheduled to receive a tetanus booster vaccination within one month before or after the influenza vaccination, response to tetanus will also be quantified. This sample will be collected during the same phlebotomy as the influenza sample. In some cases, a blood sample was stored prior to rituximab treatment and will be used for baseline assessment. The primary and secondary objectives for this study are as follows:

Primary:

* To determine the portion of patients who will respond adequately to influenza vaccination, with adequacy defined as a titer greater than 1:32 for each strain of virus in the vaccine, measured 4-8 weeks after administration of the vaccine OR greater than a four-fold increase in titers measured 4-8 weeks after administration of the vaccine

Secondary Objectives:

* To evaluate the ability to mount a response to the influenza vaccine, with response defined as any increase in influenza antibody titer for each strain of virus between samples before and 4-8 weeks after vaccination.
* To evaluate the ability to mount an adequate response to tetanus toxoid, with adequacy defined as in the primary objective.
* To evaluate the ability to mount a response to tetanus toxoid, with response defined as above.
* To compare response to influenza vaccination received less than one year after rituximab and greater than one year after rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Previously or currently enrolled in parent study, see CHB 02-12-160

Exclusion Criteria:

* Baseline immunodeficiency (i.e. DiGeorge syndrome, Common Variable Immunodeficiency)
* Contraindications for influenza vaccine, including: hypersensitivity to egg products; history of Guillain-Barre syndrome; history of adverse reaction to flu vaccine
* Contraindications for tetanus toxoid, including: hypersensitivity to prior tetanus vaccination; concurrent moderate to severe illness
* Subjects meeting any of the following criteria will be temporarily excluded from the study: high-dose corticosteroid therapy (5-30 mg/kg/day) during the 24 hours immediately prior to the vaccine; IVIG (intravenous immunoglobulin) within 4 months prior to vaccine; platelet count of less than 20,000/ml within one month of vaccination with evidence of grade II or higher skin bleeding, assessed at vaccine administration

Ages: 18 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2004-10; Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
The number of patients with a titer greater than 1:32 OR greater than 4-fold increase in titer for each strain of virus in the influenza vaccine at 4-8 weeks after vaccination

SECONDARY OUTCOMES:
The number of patients with any increase in titer for each strain of virus in the influenza vaccine at 4-8 weeks after vaccination
The number of patients with a titer greater than 1:32 OR greater than 4-fold increase in titer for each strain of virus in the tetanus vaccine at 4-8 weeks after vaccination
The number of patients with any increase in titer for each strain of virus in the tetanus vaccine at 4-8 weeks after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Ellis J Neufeld, MD, PhD, Principal Investigator — Boston Children's Hospital
Locations (3):
- United States (3):
  - University of California, Los Angeles, Los Angeles, California
  - Emory University School of Medicine, Atlanta, Georgia
  - Children's Hospital, Boston, Massachusetts